CLINICAL TRIAL: NCT07232225
Title: OCT-Based Screening for Early Retinal Changes in Asymptomatic Diabetic Patients
Acronym: DREAM-OCT
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abanoub Rafaat Marsis Rizkallah, Resident Physician / Master's Candidate, Ophthalmology Department, Assiut University
Other Study IDs: OCT DME
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asymptomatic Diabetic Patients: Patients diagnosed with Type 1or Type 2 Diabetes Mellitus for at least 6 months,BCVA 6/6, no visual symptoms, clear ocular media, no significant changes on fundus examination, and fulfilling all inclusion/exclusion criteria.
  (Total n=56)
  Interventions: Diagnostic Test: Spectral Domain OCT Imaging
- Healthy Control Subjects: Age-matched healthy subjects with no history of diabetes mellitus, BCVA 6/6, no visual symptoms, and fulfilling all study inclusion/exclusion criteria except for the diagnosis of diabetes. (Total n=56)
  Interventions: Diagnostic Test: Spectral Domain OCT Imaging

INTERVENTIONS:
Diagnostic Test: Spectral Domain OCT Imaging — Non-invasive spectral domain optical coherence tomography(SD-0CT) imaging using a NIDEK RS-330 device to measure central macular , parafoveal, and perifoveal thickness and to assess the structural integrity and layers of the retina. This is a diagnostic procedure performed for observation only.

SUMMARY:
The goal of this observational study is to detect early retinal changes in people with diabetes who do not have visual symptoms. The study will use Optical Coherence Tomography (OCT) and fundus examination to screen for early retinal involvement in diabetic patients.

The main questions this study aims to answer are:

Can OCT detect early retinal changes before symptoms appear in people with diabetes?

Is fundus examination useful for identifying early diabetic retinal changes?

Participants will undergo a comprehensive eye examination, including OCT macular scans and fundus examination, at Assiut Ophthalmology Hospital. No treatment or invasive procedures will be performed as part of this study.

The collected data will help improve early detection and prevention of diabetic retinal complications.

DETAILED DESCRIPTION:
Diabetic retinopathy is a leading cause of vision impairment worldwide. Even in the absence of visual symptoms, patients with diabetes may already have early structural retinal changes that can be detected only with advanced imaging. Identifying these changes at an early stage is essential to prevent progression to vision-threatening complications.

This observational cross-sectional study aims to evaluate the role of Optical Coherence Tomography (OCT) and fundus examination in detecting early retinal changes among diabetic patients with no visual complaints. The study will be conducted at the Ophthalmology Department, Assiut University Hospitals, Egypt.

Eligible participants will include individuals with a confirmed diagnosis of type 1 or type 2 diabetes mellitus for at least six months, best-corrected visual acuity of 6/6, clear ocular media, and no clinical evidence of retinal disease. A control group of healthy subjects with normal ocular findings will also be included for comparison.

All participants will undergo a complete ophthalmic assessment that includes:

Medical and ocular history, including diabetes duration and systemic status.

Visual acuity measurement (uncorrected and best-corrected) using the Snellen chart.

Anterior segment evaluation by slit-lamp biomicroscopy.

Fundus examination using slit-lamp biomicroscopy.

Spectral-domain OCT macular scanning (NIDEK RS-330, Japan) for assessment of macular thickness and retinal layer structure.

Data will be analyzed using SPSS software (Version 16). Quantitative variables will be expressed as mean ± standard deviation and compared using appropriate statistical tests. Correlations between OCT parameters, disease duration, and HbA1c levels will be evaluated.

The study is non-interventional and poses no significant risk to participants, as it involves only routine, non-invasive ophthalmic imaging. The findings are expected to improve early detection strategies for diabetic retinal changes and support the use of OCT and fundus examination as effective screening tools in routine diabetic eye care.

The estimated sample size will include approximately 112 participants (56 diabetic patients and 56 healthy controls).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of type 1 or type 2 diabetes mellitus for at least 6 months
* Best-corrected visual acuity (BCVA) of 6/6 using Snellen chart
* No visual symptoms (no blurred vision or metamorphopsia)
* Clear ocular media allowing high-quality OCT imaging
* No significant abnormalities on fundus examination
* Intraocular pressure (IOP) below 21 mmHg
* Willing and able to provide written informed consent

Exclusion Criteria:

* History of previous macular disease or treatment (laser photocoagulation or intravitreal injection)
* Media opacity that prevents adequate OCT imaging (e.g., dense cataract, corneal opacity)
* Presence of other retinal diseases (e.g., age-related macular degeneration, retinal vein occlusion)
* Systemic or neurological diseases that affect the retina or visual pathway
* Uncooperative participants or those who decline to give consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the Ophthalmology Department at Assiut Ophthalmology Hospital, Egypt.
  The study will include two groups:
  Group 1: Patients diagnosed with type 1 or type 2 diabetes mellitus for at least 6 months, without visual symptoms and with normal fundus examination findings.
  Group 2: Age- and sex-matched healthy individuals without diabetes, serving as controls.
  All participants will undergo a comprehensive ophthalmic examination, including best-corrected visual acuity testing, intraocular pressure measurement, fundus examination and spectral-domain optical coherence tomography (SD-OCT) imaging for retinal evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of retinal thickness parameters between diabetic patients and healthy controls | Baseline ( single assessment at the time of enrollment )
  Measurement of central macular thickness (CMT), parafoveal, and perifoveal thickness (in micrometers) using Spectral Domain OCT and assessment of retinal layer structural integrity abnormalities (e.g., intraretinal fluid or hard exudates).

SECONDARY OUTCOMES:
Correlation between OCT changes and duration of diabetes/HbA1c level | Baseline ( single assessment at the time of enrollment )
  Assessment of the statistical correlation between the measured retinal thickness parameters (CMT, parafoveal, and perifoveal thickness) and clinical variables, specifically the duration of diabetes mellitus (in years) and the latest recorded HbA1c level (in %).

REFERENCES:
- [Result] Gu Q, Pan T, Cheng R, Huang J, Zhang K, Zhang J, Yang Y, Cheng P, Liu Q, Shen H. Macular vascular and photoreceptor changes for diabetic macular edema at early stage. Sci Rep. 2024 Sep 4;14(1):20544. doi: 10.1038/s41598-024-71286-6. PMID 39232012
- [Result] Kim JT, Lee MW. Longitudinal changes in each retinal layer thickness in patients with moderate or more severe diabetic retinopathy taking calcium dobesilate. PLoS One. 2025 Jun 4;20(6):e0325655. doi: 10.1371/journal.pone.0325655. eCollection 2025. PMID 40465771
- [Result] Aldakhil S, Challa N, Alhoshan SA, Abohaimed F, Alnasser BN, Almuhawas HA, AlObaisi S, Alrasheed SH. Quantitative Analysis of Early Retinal Changes and OCT Parameters in Diabetic Subjects with and Without Retinopathy. Diagnostics (Basel). 2025 Feb 13;15(4):451. doi: 10.3390/diagnostics15040451. PMID 40002602
- [Result] Kalaw FGP, Sharma P, Walker E, Borooah S. Differences in macular thickness associated with peripheral retinal vessel whitening in diabetic patients. Sci Rep. 2024 Aug 27;14(1):19881. doi: 10.1038/s41598-024-68839-0. PMID 39191790
- [Result] Endo H, Kase S, Tanaka H, Takahashi M, Katsuta S, Suzuki Y, Fujii M, Ishida S, Kase M. Factors based on optical coherence tomography correlated with vision impairment in diabetic patients. Sci Rep. 2021 Feb 4;11(1):3004. doi: 10.1038/s41598-021-82334-w. PMID 33542264
- [Result] Shah J, Tan B, Wong D, Abdul Gani NFB, Hu Q, Liu X, Chua J. Evaluation of thickness of individual macular retinal layers in diabetic eyes from optical coherence tomography. Sci Rep. 2024 Aug 2;14(1):17909. doi: 10.1038/s41598-024-68552-y. PMID 39095380